CLINICAL TRIAL: NCT00676975
Title: Dose Escalation Trial of Traditional Chinese Medicine for Irritable Bowel Syndrome(TCM- IBS)
Brief Title: The Efficacy of Tradition Chinese Medicine in Patients With Irritable Bowel Syndrome
Acronym: TCM-IBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Maryland (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Francis KL Chan, professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM-IBS; 1U19AT003266-01 (NIH)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel disease; Traditional Chinese Medicine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Chinese Medicine (Active Comparator): Traditional Chinese Medicine 17g herbal extract
  Interventions: Drug: Traditional Chinese Medicine
- Traditional Chinese Medicine Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Traditional Chinese Medicine Placebo

INTERVENTIONS:
Drug: Traditional Chinese Medicine — A herbal extract 17g once daily for 8 weeks for lower dosage, and 34g for higher dosage.
  The 20-herb formulation are Agastache rugosa,Fraxinus rhynchophylla, Angelica dahurica,Glycyrrhiza uralensis, Artemisia capillaris, Magnolia officinalis, Atractylodes macrocephala,Paeonia lactiflora, Aucklandia lappa, Plantago asiatica,Bupleurum chinense, Phellodendron amurense, Citrus reticulate, Poria cocos, Codonopsis pilosula, Saposhnikovia diraricata, Coix lacryma-jobi, Schisandra chinensis, Coptis chinensis, Zingiber officinale
  Arms: Traditional Chinese Medicine
Drug: Traditional Chinese Medicine Placebo — Placebo once daily for 8 weeks
  Arms: Traditional Chinese Medicine Placebo

SUMMARY:
To test the efficacy of Traditional Chinese Medicine in relieving symptoms and change of quality of life of patients with Irritable Bowel Syndrome.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS), characterized by abdominal pain/discomfort and disturbed bowel frequency, is a common functional bowel disorder that accounts for a substantial proportion of patients seen in primary care and secondary referral centers. The impact on patients' quality of life and the economic burden on the community are considerable. However, the outcome of conventional Western medicine in treating IBS has been disappointing. Several potential new therapeutic agents have been withdrawn because of serious adverse events. Traditional Chinese medicine (TCM) has been used in the treatment of IBS for centuries in Asian countries but scientific evaluation of its therapeutic function is scarce. A methodologically strong trial of a 20-herb formula has shown significant benefit for IBS patients. However, the herbal formulation was inadequately characterized and defined for repeated clinical studies.

Subsequent to complete chemical characterization, a randomized, placebo-controlled, double-blind, phase II dose-escalation clinical trial will be conducted to find an optimally safe and efficacious dosage of this standardized 20-herb preparation in 104 patients aged 18 to 75 with all types of IBS. At each of two dosage levels, 52 participants will be randomized to treatment for 8 weeks with the herbal formula or placebo in a 1:1 allocation ratio, and will be assessed at baseline, weeks 0, 2, 4, 8, and 12 for the clinically important and reliable outcome of patient reported global symptom improvement. At the conclusion of the 1st dosage level, safety will be assessed prior to using the higher dosage in a new cohort of participants. We also will assess individual IBS symptoms, nature, severity, duration, and frequency of adverse events, quality of life, concurrent IBS medications and health care utilization, and will perform blood tests for safety purposes. Adherence to study medication will be verified by dose counts. Results of this dose-ranging study will help to identify the optimal dosage of the herbal formula to be used in future randomized placebo-controlled trials and in head-to-head comparisons with conventional pharmaceuticals.

ELIGIBILITY:
Inclusion Criteria:

* All IBS patients attending the Gastroenterology Clinic of the Prince of Wales Hospital of Hong Kong.
* Age 18-75 inclusive
* IBS diagnosed by Rome III criteria:

  * Recurrent abdominal pain or discomfort at least three days per month in the previous three months
  * Symptom onset at least six months prior to diagnosis
  * Pain or discomfort associated with two or more of the following:

    1. Improvement with defecation
    2. Onset associated with a change in frequency of stool
    3. Onset associated with a change in form (appearance) of stool
* Normal colonic evaluation (colonoscopy or barium enema) in past 5 years
* No "global symptom improvement" as rated by patients (see below) at baseline and during the two-week run-in period
* Normal full blood count, liver function test and renal function test.
* Informed written consent for participation into study.
* Ethical approval will be obtained from the Joint CUHK-NTEC Clinical Research Ethics Committee as well as the IRB of UMB.

Exclusion Criteria:

* Past or present history of organic disease of gastrointestinal tract (e.g. colorectal cancer, advanced colonic polyp, celiac disease, inflammatory bowel disease, peptic ulcer and previous gastrointestinal surgery). (Note: those with polyps removed during colonoscopy can be included, as long as no known polyps remained).
* Systemic diseases that cause diarrhea or constipation (e.g. thyroid disease, diabetic neuropathy)
* Lactose intolerance
* Severe liver diseases (e.g. cirrhosis, chronic active hepatitis)
* Renal impairment (serum creatinine level > 150mmol/L)
* Women who are pregnant, lactating or not practicing proper contraception
* Known hypersensitivity to herbal medicine
* Concommitant use of prescription antidepressant medication.
* Current alcoholism and drug abuse
* Current psychiatric illness or dementia
* Fever or severe illness at baseline (week 0).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-05-26 (Actual); Primary Completion 2010-12-30 (Actual); Study Completion 2011-08-30 (Actual)

PRIMARY OUTCOMES:
Patient reported global symptom improvement, based on this question: "Have you had adequate relief of your symptoms over the last two weeks"? (yes/no) | 12 weeks

SECONDARY OUTCOMES:
Bowel Symptom Scale (BSS): to assess changes in individual IBS and global IBS symptoms. QoL assessment:one disease-specific (IBS-QoL) and one generic (SF-36), will be used. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francis KL Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Li Ka Shing Specialist Clinic, Prince of Wales Hospital, Hong Kong (sar), China

IPD SHARING:
Plan to Share IPD: No